CLINICAL TRIAL: NCT01306708
Title: Comparative Study Between Amitriptyline Regarding Nimesulide Associated to Nervous Blockade in the Acute Treatment of Idiopathic Adhesive Capsulitis
Brief Title: Amitriptyline Regarding Nimesulide in Acute Idiopathic Adhesive Capsulitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidade do Sul de Santa Catarina (Other Government)
Responsible Party: Principal Investigator, Anna Paula Piovezan, Dra Anna Paula Piovezan, Universidade do Sul de Santa Catarina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10.023.4.01.III; 10.023.4.01 III (Other: Universidade do Sul de Santa Catarina)
Record Dates: First submitted 2011-03-01; First posted 2011-03-02 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2011-09

CONDITIONS: Adhesive Capsulitis
Keywords: Adhesive Capsulitis; Shoulder; SPADI
MeSH Terms: conditions — Bursitis | interventions — Amitriptyline

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- nimesulide (Active Comparator): Nerve suprascapular blockade with local anaesthetic agent (novabupivacaine 0.25%, 10 ml, once per week) + oral non-steroidal anti-inflammatory (nimesulide 100 mg, twice per day, for 14 days);
  Interventions: Drug: amitriptyline

INTERVENTIONS:
Drug: amitriptyline — Nerve suprascapular blockade with local anaesthetic agent (novabupivacaine 0.25%, 10 ml, once per week) + oral tricyclic antidepressant (amitriptyline 25 mg, twice per day, for 14 days);

SUMMARY:
The adhesive capsulitis is a disease of the shoulder characterized by pain and limitation of movement amplitude. It is defined as for etiology, having discordant theories that related it to an inflammatory condition or to an algoneurodystrophy process. There is not yet a consensus about the best option of treatment. The non-steroidal anti-inflammatories have analgesic and anti-inflammatory activity, where the mechanism of action is the inhibition of prostaglandin synthesis. The antidepressants have been increasingly used in the control of chronic pain and the major action mechanism to have the analgesic effect seems to be based on inhibition of neurotransmitters reuptake noradrenaline and/or serotonin) in nerve cell endings. Literature studies associate the practice of the nerve suprascapular blockade with anaesthetics to good results of clinical improvement of the pain, however, so far, no clinical studies comparing the efficacy of the non-steroidal antiinflammatories or tricyclic antidepressants to nervous blockage were registered in the acute treatment of adhesive capsulitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical diagnostic of adhesive capsulitis, phase II, presenting shoulder pain,
* Limitation of anterior elevation for up to 130 degrees,
* Intact rotator cuff to magnetic resonance,
* Minimum loss of 50% of external rotation when compared to the contralateral side.
* Patients' acceptance of take part in the study after signing the FCCT.

Exclusion Criteria:

* Incapacity to fill the evaluation instrument;
* Contraindication to the use of local anaesthetics, non-steroidal anti-inflammatories or tricyclic antidepressants.
* Pregnancy and breastfeeding.
* Not follow the orientations during treatment on the weeks included in the study, such as, using other anaesthetics or procedures for the relief of pain in this period.
* Lesion of the rotator cuff, infection and others arthropathies.
* Inability to fill a protocol.
* Previous surgery on the shoulder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2011-02; Primary Completion 2011-07 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Pain and disability of the shoulder | Days 0 and 14 after treatment begining
  Pain and disability of the shoulder, measured by the use of SPADI questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Anna P Piovezan, Doctor, Principal Investigator — Universidade do Sul de Santa Catarina
Locations (1):
- Universidade do Sul de Santa Catarina, Tubarão, Santa Catarina, Brazil